CLINICAL TRIAL: NCT05735522
Title: Randomized, Sham-controlled Study on the Effectiveness of Magnetic Stimulation in the Treatment of Female Urgency Urinary Incontinence.
Brief Title: Effectiveness of Magnetic Stimulation in the Treatment of Female UUI.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Principal Investigator, David Lukanovic, asist. dr., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMCL-UUI
Record Dates: First submitted 2023-01-19; First posted 2023-02-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Urge; Pelvic Floor Disorders
Keywords: urgency urinary incontinence; urinary incontinence; magnetic stimulation; urinary urgency
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge; Pelvic Floor Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): We are using an extracorporeal magnetic stimulation chair with two magnetic stimulators, one under the seat and one in the backrest, that generate the magnetic field. The treatment lasts for 30 minutes and has 5 steps. Each step has a defined duration and a defined frequency of magnetic field pulsations. In each step, it is also defined, which of the magnetic field generators are working. The pulsations last for 6 seconds followed by 6 seconds of rest.
  Step 1: 10Hz, 7 minutes, 6 seconds on, 6 seconds off, both stimulators generate the magnetic field. Step 2: 10Hz, 4 minutes, the stimulator under the seat generates the magnetic field. Step 3: 10Hz, 7 minutes, the stimulator in the backrest generates the magnetic field. Step 4: 30Hz, 10 minutes, both stimulators generate the magnetic field. Step 5: After 5 minutes, both stimulators generate the magnetic field.
  During the treatment, we adjusted the magnetic field density. It varied from 2-100%. The maximum was 3 Teslas.
  Interventions: Device: Extracorporeal magnetic stimulation
- Sham group (Sham Comparator): We are using extracorporeal magnetic stimulation, a chair with two magnetic stimulators, one under the seat and one in the backrest, that generate the magnetic field. The treatment lasts for 30 minutes and has 5 steps. We used the same program as in the active group with the difference that the magnetic field density was always at 2% so the effects of the pulsating are negligible.
  Interventions: Other: Sham

INTERVENTIONS:
Device: Extracorporeal magnetic stimulation — Extracorporeal magnetic stimulation is a technique based on Faraday's law of magnetic induction, approved by the United States Food and Drug Administration in 1998, for conservative treatment of urinary incontinence. It generates electrical activity, which induces controlled depolarization of the nerves, resulting in pelvic muscle contraction and sacral S2-S4 roots neuromodulation. The patient seats in the chair fully clothed.
  Arms: Active group
Other: Sham — The same chair as is used in the active group with the magnetic field density at the lower 2% resulting in negligible efficacy.
  Arms: Sham group

SUMMARY:
Urinary incontinence is becoming an increasingly common health, social and economic problem. The prevalence of urinary incontinence is estimated at 55% of the entire female population. Urgency urinary incontinence (UUI) is the least common subtype of urinary incontinence but has debilitating symptoms that lead to a decrease in quality of life. Ultimately, the urogynegology field does not have many successful types of treatments for this specific subtype. Extracorporeal magnetic stimulation of the pelvic floor is a type of conservative management that produces a magnetic field, which induces controlled depolarization of the nerves, resulting in pelvic muscle contraction and sacral S2-S4 roots neuromodulation. Therefore, it relieves symptoms of UUI and improves quality of life.

There was no randomized, sham-controlled study published that researched the effectiveness of magnetic stimulation in the treatment of UUI that evaluated the success with subjective and objective methods, such as urodynamic studies.

The aim of this study was to assess the efficacy of magnetic stimulation in the treatment of urgency urinary incontinence.

DETAILED DESCRIPTION:
RATIONALE: The FDA approved extracorporeal magnetic stimulation as a form of conservative treatment of urinary incontinence in 1998. Since then, the studies focused mainly on magnetic stimulation's effectiveness in treating stress urinary incontinence. There are five studies that assessed the efficacy of magnetic stimulation in the treatment of urgency urinary incontinence. Only one was randomized and sham-controlled, others were not. Three studies used urodynamic studies to assess the effectiveness of magnetic stimulation treatment, but those studies were not randomized or sham-controlled. The EAU guidelines, therefore, do not recommend extracorporeal magnetic stimulation as a treatment option for urinary incontinence for the lack of evidence.

AIM OF THE STUDY: The study will evaluate the efficacy of magnetic stimulation as a type of conservative treatment in patients with urgency urinary incontinence. After evaluating previously conducted studies, the investigators decided to conduct the first randomized, sham-controlled study that evaluated the effectiveness of magnetic stimulation as a treatment for urgency urinary incontinence with subjective and objective measures.

METHODS: the study will be randomized and sham controlled with 40 enrolled patients. The patients will be allocated in the active or sham arm in a ratio of 2:1. The patients will be recruited from the UMC Ljubljana outpatient urogynecologic clinic. All eligible patients will be invited to participate in our study by phone.

STATISTICAL ANALYSES: The results will be analysed with the Kolmogorov-Smirnov test and two-way ANOVA with repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* urgency urinary incontinence proved by urodynamic studies
* 18 years of age

Exclusion Criteria:

* pregnancy
* cystitis or other active infections
* stress or mixed urinary incontinence
* prolapse of pelvic organs with POP-Q score greated than 2
* fecal incontinence
* severe medical conditions (e.g. active treatment of cancer)
* connective tissue disease
* neurologic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Change in the ICIQ-UI SF score | Before the treatment and immediately after the treatment, 3 months after the treatment, 6 months after the treatment and 12 months after the treatment.
  Difference in the score of the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) questionnaire. The scoring scale is 0-21 points. Lower score means better outcome.
Change in voiding diary 1 | Before the treatment and immediately after the treatment, 3 months after the treatment, 6 months after the treatment and 12 months after the treatment.
  Difference in the mean voided volume. Higher mean voided volume means better outcome.
Change in voiding diary 2 | Before the treatment and immediately after the treatment, 3 months after the treatment, 6 months after the treatment and 12 months after the treatment.
  Difference in the mean number of incontinence episodes. Lower number of incontinence episodes means better outcome.
Change in voiding diary 3 | Before the treatment and immediately after the treatment, 3 months after the treatment, 6 months after the treatment and 12 months after the treatment.
  Difference in the mean number of micturitions. Lower number of micturitions means better outcome.
Change in urodynamic studies 1 | Before the treatment and 3 months after the treatment.
  Difference in the volume at first desire to void. Higher volume means better outcome.
Change in urodynamic studies 2 | Before the treatment and 3 months after the treatment.
  Difference in the maximum cystometric capacity. Higher volume means better outcome.

SECONDARY OUTCOMES:
Change in UDI-6 score | Before the treatment and immediately after the treatment, 3 months after the treatment, 6 months after the treatment and 12 months after the treatment.
  Difference in the score of the Urinary Distress Inventory Short Form (UDI-6) questionnaire. Score values go from 0 to 100. Lower score means better outcome.
Change in IIQ-7 score | Before the treatment and immediately after the treatment, 3 months after the treatment, 6 months after the treatment and 12 months after the treatment.
  Difference in the score of the Incontinence Impact questionnaire Short Form (IIQ-7) questionnaire. Scores go from 0 to 100 with lower score meaning better outcome.
Change in PISQ-12 score | Before the treatment and immediately after the treatment, 3 months after the treatment, 6 months after the treatment and 12 months after the treatment.
  Difference in the score of The Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12). Scores go from 0 to 48 with higher score meaning better outcome.
Change in King's Health questionnaire | Before the treatment and immediately after the treatment, 3 months after the treatment, 6 months after the treatment and 12 months after the treatment.
  Difference in the score of the King's health questionnaire. Scores go from 0 to 100. With lower score meaning better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Adolf Lukanović, MD, PhD, Principal Investigator — Department of Gynecology, Division of Gynecology and Obstetrics, Ljubljana University Medical Center
Locations (1):
- Department of Gynecology, Division of Gynecology and Obstetrics, Ljubljana University Medical Center, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in UUI.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 20 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of the principal investigator.For more information or to submit a request, please contact david.lukanovic@kclj.si

REFERENCES:
- [Background] Lukanovic D, Kunic T, Batkoska M, Matjasic M, Barbic M. Effectiveness of Magnetic Stimulation in the Treatment of Urinary Incontinence: A Systematic Review and Results of Our Study. J Clin Med. 2021 Nov 8;10(21):5210. doi: 10.3390/jcm10215210. PMID 34768730
- [Background] He Q, Xiao K, Peng L, Lai J, Li H, Luo D, Wang K. An Effective Meta-analysis of Magnetic Stimulation Therapy for Urinary Incontinence. Sci Rep. 2019 Jun 24;9(1):9077. doi: 10.1038/s41598-019-45330-9. PMID 31235706
- [Background] Yamanishi T, Homma Y, Nishizawa O, Yasuda K, Yokoyama O; SMN-X Study Group. Multicenter, randomized, sham-controlled study on the efficacy of magnetic stimulation for women with urgency urinary incontinence. Int J Urol. 2014 Apr;21(4):395-400. doi: 10.1111/iju.12289. Epub 2013 Oct 14. PMID 24118165